CLINICAL TRIAL: NCT02309931
Title: Randomized Clinical Trial Comparing Isoperistaltic Versus Antiperistaltic Side to Side Anastomosis After Right Laparoscopic Hemicolectomy for Cancer.
Brief Title: ISOperistaltic Versus ANTIperistaltic Anastomosis After Laparoscopic Right Colectomy for Cancer
Acronym: ISOVANTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Jesus Abrisqueta Carrion, Ph D, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCR-HCUVA-2014-01
Record Dates: First submitted 2014-11-28; First posted 2014-12-05 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Primary Malignant Neoplasm of Ascending Colon
Keywords: Right hemicolectomy; Side-to-side anastomosis; Orocecal time; Antipersitaltic; Isoperistaltic; Laparoscopic colectomy; Right laparoscopic hemicolectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoperistaltic anastomosis (Active Comparator): Patients with right colon cancer who undergo a right laparoscopic hemicolectomy and a isoperistaltic side-to-side ileocecal anastomosis
  Interventions: Procedure: isoperistaltic side-to-side ileocecal anastomosis
- Antiperistaltic anastomosis (Active Comparator): Patients with right colon cancer who undergo a right laparoscopic hemicolectomy and a antiperistaltic side-to-side ileocecal anastomosis
  Interventions: Procedure: antiperistaltic side-to-side ileocecal anastomosis

INTERVENTIONS:
Procedure: antiperistaltic side-to-side ileocecal anastomosis — Right laparoscopic hemicolectomy + antiperistaltic side-to-side ileocecal anastomosis
  Arms: Antiperistaltic anastomosis
Procedure: isoperistaltic side-to-side ileocecal anastomosis — Right laparoscopic hemicolectomy+isoperistaltic side-to-side ileocecal anastomosis
  Arms: Isoperistaltic anastomosis

SUMMARY:
The study will provide a precise control compared to the two interventions (iso vs antiperistaltic anastomoses) with thorough measurements of the postoperative variables and complications to improve the evaluation of the surgical technique. It will also enable an evaluation of the quality of life after the procedures.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given informed consent to participate
* No surgery contraindications
* Elective surgery
* No pregnancy or nursery during the study
* Older than 18 years
* Complete preoperative cancer staging
* Tumour characteristics:

  * Cecum, ascending, hepatic angle or transverse colon tumour confirmed by endoscopic biopsy
  * Radiologically resectable tumours
  * Absence of vascular, nervous or bone infiltration
  * T4 stages with near organ infiltration
  * Absence of peritoneal carcinomatosis
  * Absence of respiratory pathology that prevents for doing hydrogen breath test

Exclusion Criteria:

* Pregnancy
* Intestinal bowel disease like Crohn's disease or ulcerative colitis.
* Metastatic bone illness
* Previous abdominal surgery with bowel resection
* Malabsorption syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
postoperative complications | within the first 30 days up to one year after surgery
  Number of patients with postoperative complications and grade of Clavien-Dindo

SECONDARY OUTCOMES:
Operating time | During surgery
Anastomosis time | From the enteromy to its closure.
Hospital length of say | participants will be followed for the duration of hospital stay, an expected average of 4 days
first tolerance day | participants will be followed for the duration of hospital stay, an expected average of 4 days
  First day taking liquids without vomits or abdominal distension
first flatus day | participants will be followed for the duration of hospital stay, an expected average of 4 days
first faeces day | participants will be followed for the duration of hospital stay, an expected average of 4 days
Orocecal transit | up to one year
  Using hydrogen breath test curves. preoperative, at day 2 postoperative, 1 month, 6 months and 1 year.
Gastrointestinal life quality | up to one year
  Using gastrointestinal quality life index questionnaire. preoperative, 1 month, 6 months and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Lujan, Ph D, Study Director — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Universitario Virgen de La Arrixaca, Murcia, Spain

REFERENCES:
- [Derived] Ibanez N, Abrisqueta J, Lujan J, Hernandez Q, Rufete MD, Parrilla P. Isoperistaltic versus antiperistaltic ileocolic anastomosis. Does it really matter? Results from a randomised clinical trial (ISOVANTI). Surg Endosc. 2019 Sep;33(9):2850-2857. doi: 10.1007/s00464-018-6580-7. Epub 2018 Nov 13. PMID 30426254
- [Derived] Ibanez N, Abrisqueta J, Lujan J, Hernandez Q, Parrilla P. Isoperistaltic versus antiperistaltic side-to-side anastomosis after right laparoscopic hemicolectomy for cancer (ISOVANTI) trial: study protocol for a randomised clinical trial. Int J Colorectal Dis. 2017 Sep;32(9):1349-1356. doi: 10.1007/s00384-017-2840-6. Epub 2017 Jun 21. PMID 28634703